CLINICAL TRIAL: NCT04198051
Title: The Clinical Study of Adjuvant Chemotherapy on Intestinal and Urethral Flora in Patients With Gastric and Colon Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Dalian Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PJ-KY-2019-101
Record Dates: First submitted 2019-12-03; First posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-09

CONDITIONS: Gastric Cancer; Colon Cancer
MeSH Terms: conditions — Stomach Neoplasms; Colonic Neoplasms | interventions — Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental)
  Interventions: Drug: adjuvant chemotherapy

INTERVENTIONS:
Drug: adjuvant chemotherapy — Form、dosage and frequency： Gastric cancer was given the SOX regimen (oxaliplatin + tegafur regimen,oxaliplatin 130mg/m2 intravenous infusion, the 1st day; tegafur 80mg/ m2/d orally Bid, the 1st to 14th day, every 21 days is one cycle) or XELOX regimen (oxaliplatin + capecitabine regimen，oxaliplatin 130mg/m2 intravenous infusion, the 1st day; capecitabine 1000mg/m2/d orally Bid, the 1st to 14th day, every 21 days is one cycle).
  Colon cancer was given the XELOX regimen (the dosage、frequency and administration are the same as the gastric cancer) or FOLFOX regimen (oxaliplatin + calcium folinate + fluorouracil regimen，oxaliplatin 85mg/m2 intravenous infusion, the 1st day; calcium folinate 400 mg/m2 intravenous infusion, the 1st day; fluorouracil 400 mg/m2 intravenous infusion, the 1st day, then 1200 mg/m2/d × 2d continuous intravenous infusion，every 14 days is one cycle).
  Duration：through chemotherapy completion，about six months.

SUMMARY:
The human intestine is colonized with a complex microbial community and forms a super organism with the human body. Intestinal microorganisms include more than 1,000 kinds of bacterias, and their flora is very complex and functions are very diverse. The intestinal flora affects the body's nutrition, immunity and metabolism through interaction with the human body and the external environment, and is closely related to multiple systems. When the flora structure and function are changed, it will lead to the occurrence of various diseases or increase the risk of disease. In recent years, the role of intestinal microbes in tumorigenesis and development, as well as the role of diagnosis and treatment have been paid more and more attention. Abnormal intestinal flora can not only promote tumorigenesis, but also affect radiochemotherapy and immunotherapy effects. It is worth noting that the huge impact of the intestinal flora on immunotherapy suggests that immune checkpoint inhibitors can maximize the efficacy by protecting the balance and diversity of the intestinal microecology. Therefore, in this study, quantitative analysis of the diversity and abundance of intestinal, urinary tract flora, and urine components before and after adjuvant chemotherapy in patients with gastric and bowel cancer was performed. The link between treatment efficacy and prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years old, male or female
2. Surgery specimens were clearly diagnosed as gastric cancer and colon cancer by histopathology
3. The operation method is not limited (both laparoscopic surgery and open surgery)
4. After the perioperative period, stop using antibiotics for not less than 2 weeks
5. It is planned to receive a chemotherapy regimen with a combination of platinum and fluorouracil for a period of 21 days (gastric cancer is the SOX or XELOX regimen, and colon cancer is the XELOX or FOLFOX regimen)
6. Blood routine, biochemical and other related laboratory tests showed no obvious abnormalities
7. There are no contraindications for related adjuvant chemotherapy indications.

Exclusion Criteria:

1. Neoadjuvant treatment before gastric and bowel cancer surgery
2. Previous history: He has suffered from intestinal microecology-related diseases such as cirrhosis, ulcerative colitis, Crohn's disease, irritable bowel syndrome, and urinary system diseases
3. Before the perioperative period, because of anastomotic fistula and gastrointestinal perforation, reoperation
4. The following drugs were used within 2 weeks before enrollment:

   1. Various antibiotics, including antifungals (oral and intravenous)
   2. Probiotic preparations, various prebiotic preparations, etc c Glucocorticoids; d Take drugs known to have a significant effect on the intestinal and urethral flora within half a year (such as proton pump inhibitors, purgatives, bismuth, adsorbents, non-steroidal anti-inflammatory drugs, etc.)
5. Other situations that the researcher considers unsuitable to participate in the experiment;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-12-20 (Estimated); Primary Completion 2020-12-20 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
The change of diversity of intestinal flora in faeces during chemotherapy | The 1st day before the start of each cycle of chemotherapy, and the 1st day after the completion of each cycle of chemotherapy(each cycle is 21 days,except for the FOLFOX regimen of colon cancer is 14 days),through chemotherapy completion, six months.
The change of diversity of urethral flora in urine during chemotherapy | The 1st day before the start of each cycle of chemotherapy, and the 1st day after the completion of each cycle of chemotherapy(each cycle is 21 days,except for the FOLFOX regimen of colon cancer is 14 days),through chemotherapy completion, six months.
The change of abundance of intestinal flora in faeces during chemotherapy | The 1st day before the start of each cycle of chemotherapy, and the 1st day after the completion of each cycle of chemotherapy(each cycle is 21 days,except for the FOLFOX regimen of colon cancer is 14 days),through chemotherapy completion, six months.
The change of abundance of urethral flora in urine during chemotherapy | The 1st day before the start of each cycle of chemotherapy, and the 1st day after the completion of each cycle of chemotherapy(each cycle is 21 days,except for the FOLFOX regimen of colon cancer is 14 days),through chemotherapy completion, six months.
The change of concentration of purine metabolites in urine during chemotherapy | The 1st day before the start of each cycle of chemotherapy, and the 1st day after the completion of each cycle of chemotherapy(each cycle is 21 days,except for the FOLFOX regimen of colon cancer is 14 days),through chemotherapy completion, six months.
The change of concentration of P-hydroxyphenylalanine metabolites in urine during chemotherapy | The 1st day before the start of each cycle of chemotherapy, and the 1st day after the completion of each cycle of chemotherapy(each cycle is 21 days,except for the FOLFOX regimen of colon cancer is 14 days),through chemotherapy completion, six months.

SECONDARY OUTCOMES:
The change of the number of Gastrin in blood during chemotherapy | the 1st day before the start of each cycle of chemotherapy(each cycle is 21 days,except for the FOLFOX regimen of colon cancer is 14 days),through chemotherapy completion, 6 months.
The change of the number of CD4+T cell and CD8+T cell in blood during chemotherapy chemotherapy | the 1st day before the start of each cycle of chemotherapy(each cycle is 21 days,except for the FOLFOX regimen of colon cancer is 14 days),through chemotherapy completion, 6 months.
The change of the number of Interleukin(IL)-2,Interleukin(IL)-4,Interleukin(IL)-6, in blood during chemotherapy | the 1st day before the start of each cycle of chemotherapy(each cycle is 21 days,except for the FOLFOX regimen of colon cancer is 14 days),through chemotherapy completion, 6 months.
The change of the number of tumor necrosis factor(TNF)-α in blood during chemotherapy | the 1st day before the start of each cycle of chemotherapy(each cycle is 21 days,except for the FOLFOX regimen of colon cancer is 14 days),through chemotherapy completion, 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaonan Cui, MD,PhD, Principal Investigator — The First Affiliated Hospital of Dalian Medical University
Locations (1):
- The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided